CLINICAL TRIAL: NCT00321009
Title: A Prospective Randomized Trial Comparing Enoxaparin to Warfarin for the Prevention of LV Thrombus Formation After Anterior Wall Myocardial Infarction: A 60 Patient Pilot Study
Brief Title: LV Thrombus Pilot Study for Comparing Enoxaparin Vs. Warfarin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Rhone-Poulenc Rorer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IND 59673
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Coronary Artery Disease; Acute Myocardial Infarction
Keywords: Myocardial Infarction; Left Ventricular Mural Thrombus; Low Molecular Weight Heparin; Enoxaparin; Warfarin; Echocardiograms
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction | interventions — Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
To prospectively evaluate the utility of enoxaparin vs. oral warfarin in reduction of echocardiographic indices of LV mural thrombus. The primary outcome is the presence of LV mural thrombus at 3.5 months. The secondary outcome is cost analysis comparing the two arms.

DETAILED DESCRIPTION:
Patients with anterior Q-wave MIs and ejection fractions<=40% will be enrolled within the first 4 days of infarction. Patients will be randomized to receive either enoxaparin 1mg/kg (maximum 100mg) subcutaneously every 12 hours for one month or heparin followed by oral warfarin for 3 months.

Clinical and safety evaluations, 2-D echocardiograms at baseline and at 3.5 months and cost analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Anterior myocardial infarction with:

  1. Pathological Q-waves in at least 3 contiguous anterior precordial leads, assumed to be new
  2. CK peak>5 times the upper limit of normal with positive MB bands
* Ejection fraction <=40% or anterior dyskinesis or documented LV Thrombus
* MI onset < 7 days from randomization

Exclusion Criteria:

* Inability to give written informed consent
* Medical conditions that would prohibit discharge within 48 hours with the exception of need for anticoagulation
* Cardiogenic shock, rest angina unresponsive to medical therapy or serious ventricular arrhythmia in the 24 hours prior to randomization
* Patients scheduled for surgical procedure in the next 4 months that would prevent use of enoxaparin or warfarin
* Anemia: Baseline Hgb<=9 gm for women, <=10 gm for men or platelet count<100,000
* Renal insufficiency (creatinine >2.0 mg/dl)
* Serious liver disease as reflected by INR>1.3
* Stroke within past 6 months or a prior documented intracranial or subarachnoid hemorrhage
* Active bleeding or major surgery within 2 weeks prohibiting the use of anticoagulants
* Acute pericarditis
* Women of childbearing potential unless pregnancy test negative
* Cardiac or non-cardiac condition with expected survival< 6 months
* Severe peripheral vascular disease
* Patients who undergo cardiac surgery, including CABG, as a result of their index myocardial infarction
* Allergy to aspirin, heparin or warfarin, pork or pork products
* History of recurrent thromboembolic disease or a history of Protein C, Protein S, antithrombin III deficiency or known bleeding disorder.
* Current use of warfarin or need for chronic anticoagulation
* Current participation in other trials using investigational drugs or devices
* Prior enrollment in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2000-03; Study Completion 2004-04

PRIMARY OUTCOMES:
What is the incidence of LV mural thrombus with administration of enoxaparin vs.
warfarin at 3.5 months in patients presenting with anterior wall myocardial
infarctions.

SECONDARY OUTCOMES:
What are the associated costs and length of hospital stay after randomized to
enoxaparin vs. warfarin?

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Grines, MD, Principal Investigator — Corewell Health East
Locations (6):
- United States (6):
  - University of Colorado Health Sciences Center, Denver, Colorado
  - William Beaumont Hospital, Royal Oak, Michigan
  - St Joseph's Health Center Dept. of Cardiology, Syracuse, New York
  - LaBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Cardiovascular Associates Ltd., Virginia Beach, Virginia